CLINICAL TRIAL: NCT01472341
Title: Beta-Cell Dysfunction and Insulin Resistance Among Italian Patients With Type 2 Diabetes
Brief Title: Beta-Cell Dysfunction and Insulin Resistance Among Italian Patients With Type 2 Diabetes (MK-0000-113)
Acronym: BETADECLINE
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0000-113
Record Dates: First submitted 2011-11-11; First posted 2011-11-16 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: Participants receiving routine care under a diabetologist.

SUMMARY:
The purpose of this study is to evaluate the degree of beta-cell dysfunction among participants with type 2 diabetes and the association between beta-cell dysfunction and demographic, clinical, and treatment variables.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of type 2 diabetes mellitus by American Diabetes Association (ADA) criteria
* Oral hypoglycemic drug therapy for ≥1 year
* Continuous care at the clinic (at least 2 visits) for at least one year
* Medical records completed with a minimum core data set
* Completed consent form

Exclusion Criteria:

* Participation in a clinical trial in the previous 1 year
* Currently using insulin
* Type 1 diabetes
* Pregnancy

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants visiting a diabetologist as part of their routine care. Investigator's prescription is not influenced by the study: Investigator decides about what is the best treatment for any single participant independently of the study.
Sampling Method: Non-Probability Sample
Enrollment: 507 (Actual)
Dates: Start 2008-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0000-113&kw=0000-113&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational study was conducted at 9 outpatient diabetes clinics in Italy.
Period: Overall Study
Arm/Group | All Participants
Started | 507
Completed | 235
Not Completed | 272
Not completed — Started insulin therapy | 55
Not completed — Started therapy with a DPP-IV/GLP-1 | 92
Not completed — Withdrawal by Subject | 39
Not completed — Lost to Follow-up | 52
Not completed — Laboratory parameters unavailable | 25
Not completed — Death | 9

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 507
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209
  Male | 298

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Homeostatic Model Assessment Fasting Beta Cell Function (HOMA % B) at 4 Years
Description: HOMA is a method used to quantify insulin resistance (a condition in which natural hormone insulin becomes less effective in lowering blood sugars) and beta-cell (specialized cells in the pancreas producing insulin) function. HOMA uses fasting plasma insulin and glucose concentrations to estimate steady state pancreatic beta cell function (%B) as a percentage of a normal reference population (normal young adults). The normal reference population was set at 100%. HOMA%B was defined as 20 x fasting insulin (mU/L)/fasting glucose (mmol/L) - 3.5.
Time Frame: Baseline and 4 years
Population: Participants who had laboratory parameters at Baseline and at Year 4.
Measure: Mean (Standard Deviation); unit: Percentage of Beta Cell Function
Arm/Group | All Participants
Number analyzed (Participants) | 235
Percentage of Beta Cell Function
  HOMA-B at Baseline | 50.2 (49.1)
  HOMA-B at Year 4 | 48.3 (36.3)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p = 0.24, Multivariate regression analysis; HOMA %B was the response variable and other study parameters were independent variables

2. Primary Outcome: Change From Baseline in Proinsulin/Insulin (PI/I) Ratio at 4 Years
Description: Proinsulin is the prohormone precursor to insulin made in the beta cells of the islets of Langerhans, specialized regions of the pancreas. A raised proinsulin-to-insulin ratio due to impaired processing of proinsulin is an early marker of beta cell dysfunction. Beta-cell dysfunction was evaluated by calculating the PI/I ratio, which estimates the capacity of beta cells to convert proinsulin to insulin and may represent an acceptable method to indicate the degree of beta-cell secretion.
Time Frame: Baseline and Year 4
Population: Participants who had laboratory parameters at Baseline and at Year 4.
Measure: Mean (Standard Deviation); unit: PI/I
Arm/Group | All Participants
Number analyzed (Participants) | 235
PI/I
  PI/I at Baseline | 1.19 (1.86)
  PI/I at Year 4 | 1.61 (1.72)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p = 0.001, Multivariate regression analysis; PI/I ratio was the response variable and other study parameters were independent variables

3. Primary Outcome: Homeostatic Model Assessment Fasting Beta Cell Function (HOMA % B) According to Quartiles of Proinsulin/Insulin (PI/I) Ratio
Description: HOMA is a method used to quantify insulin resistance (a condition in which natural hormone insulin becomes less effective in lowering blood sugars) and beta-cell (specialized cells in the pancreas producing insulin) function. HOMA uses fasting plasma insulin and glucose concentrations to estimate steady state pancreatic beta cell function (%B) as a percentage of a normal reference population (normal young adults). The normal reference population was set at 100%. HOMA%B was defined as 20 x fasting insulin (mU/L)/fasting glucose (mmol/L) - 3.5. Beta-cell dysfunction was evaluated by calculating the PI/I ratio, which estimates the capacity of beta cells to convert proinsulin to insulin and may represent an acceptable method to indicate the degree of beta-cell secretion.
Time Frame: Baseline
Population: Participants with fasting plasma insulin and glucose concentration assessments at baseline.
Measure: Mean (Standard Deviation); unit: Percentage Beta Cell Function
Arm/Group | All Participants
Number analyzed (Participants) | 504
Percentage Beta Cell Function
  I. PI/PII <=0.485 | 73.4 (63.8)
  II. PI/PII 0.485 to 0.80 | 51.6 (33.2)
  III. PI/PII 0.81 to 1.355 | 37.7 (30.4)
  IV PI/PII >1.355 | 29.9 (33.4)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p < 0.0001, Multivariate regression analysis; HOMA %B was the response variable and other study parameters were independent variables

ADVERSE EVENTS:
Description: There were no plans for the systematic collection or analysis of serious adverse events (SAEs) or adverse events (AEs) in the MK-0000-113 trial. Any SAEs or AEs reported were unsolicited and non-systematically assessed.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 1/507
Other Adverse Events (participants affected / at risk) | 0/507
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=507)
Death due to parotid cancer in advanced stage [Salivary gland cancer] (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each site can publish its own results without the results of other sites after the publication of the study or after 24 months from completion of publication. The author list will be established with the participating sites before the layout of the text to be published. The company will need to evaluate all the proposed summaries, manuscripts or presentations 60 days prior to publication. The revision made by Company could be accelerated in order to satisfy the guidelines concerning publication.